CLINICAL TRIAL: NCT07103928
Title: Prison-Based HIV Partner Notification
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 2024-0926; R01MH138246 (NIH)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: HIV
Keywords: HIV; partner notification; contact tracing; sexually transmitted infections; prisons; Injection drug use
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impart Choice of APN or Self-Tell Per Partner (Experimental): Participants are assisted to identify partners whom they wish to notify and coached in how to tell their at-risk partners by the end of 6 weeks. Participants may choose per partner between sell-tell notification or having an Impart HIV-trained nurse and community outreach healthcare provider work as a team to locate, notify, and offer HIV testing to their partners.
  Interventions: Behavioral: Impart Assisted Partner Notification; Behavioral: Self-Tell Notification
- Self-Tell Notification Only Standard of Care Condition (Active Comparator): Participants are assisted to identify partners whom they wish to notify and coached in how to tell their at-risk partners by the end of 6 weeks. Participants may choose to tell their partner(s) by telephone, mail, or in-person during visitation at the jail/prison facility. They also may elect to have an Impart counselor present during in-person telling or by telephone to answer any clinical questions that the partner might have.
  Interventions: Behavioral: Self-Tell Notification

INTERVENTIONS:
Behavioral: Impart Assisted Partner Notification — Participants randomized to the Impart arm may choose per partner either a) sell-tell notification or b) having an Impart-trained APN notifier team locate, notify, and offer HIV testing to their partners without revealing the identity of who had named them. Impart notifiers initially contact named partners by telephone and identify themselves as health service providers with important information about the partner's health that needs to be shared in person. Partners who agree to meet are asked to choose a location. Notification by telephone is only delivered as a last resort when circumstances prevent in-person notification or a partner insists on learning the reason for the telephone call. Once contact is made at a private location, partners will be advised of their possible shared exposure to HIV. APN notifiers never reveal participant names or identifying information during this meeting. All notified partners are offered immediate HIV testing and treatment referral, if HIV-positive.
  Other Names: HIV partner notification; Provider-assisted partner notification
  Arms: Impart Choice of APN or Self-Tell Per Partner
Behavioral: Self-Tell Notification — Participants who wish to self-notify one or more partners are coached to do so either in person or by telephone. APN counselors confirm the names of partners for whom participants provide contact information before giving the phone to the participant to explain the reason for the call: "I want to speak with you because I was diagnosed with HIV and I believe we shared an exposure." Alternately, participants who wish to notify partners in person are coached to inform partners that they have a serious health matter that they wish to discuss, and ask the partner to visit them in jail/prison. Either way, the APN counselor is present to record the names of partners whom participants self-notify, and offers to speak with the partner immediately afterwards to answer their questions about HIV and to provide information about HIV testing and contact information should the partner wish to contact an HIV provider on their own to learn more about HIV testing or to schedule an HIV test.

SUMMARY:
Assisted partner notification (APN) is a voluntary and confidential process that utilizes specially-trained health workers to encourage and assist people diagnosed with HIV to inform their sex and drug use partners about possible shared exposure to HIV. With APN, partners who have come in contact with HIV are notified about exposure and given information to protect themselves from contracting HIV in the future or to begin treatment, if needed.

This study compares two types of HIV partner notification. Incarcerated men with HIV will be recruited as "index participants". Participants in both groups will be encouraged to notify sex and needle-sharing partners with whom they may have shared an HIV exposure before incarceration. All participants have the option to self-notify partners during a prison visitation or telephone call. In addition, participants randomized to an APN Choice group also can opt for anonymous notification by specially-trained APN notifiers that includes contact tracing if needed. As outcomes, we will compare the number of partners in each condition who are notified, HIV tested, diagnosed, and linked to HIV treatment. The study will show if prison-based APN is successful in reaching partners for HIV testing.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of Impart, an assisted partner notification (APN) intervention that was developed to increase HIV testing and referral into treatment among the sex and drug use partners of incarcerated people with HIV. Incarcerated people with HIV are assigned randomly to one of two groups. Participants assigned to the Impart Choice condition may choose to inform partners themselves by telephone or in person or they may ask specially-trained nurses and outreach workers to confidentially notify partners and to offer partners HIV testing. Meanwhile, participants assigned to the Standard of Care Self-Tell Notification Only condition will be encouraged to tell their partner(s) themselves, either by phone or in person during a prison visitation. As outcomes, we will compare after six weeks the number of partners in each condition who are notified, HIV tested, diagnosed, and linked to confirmatory HIV testing and treatment After 6 weeks, we will offer outreach-assisted partner notification to any participant who was randomized to or initially chose to notify their partners themselves. Results from the study will provide evidence as to the use of prison-based APN in making partner notification desirable and acceptable to people in prison while also reducing barriers to partner notification and HIV testing for their partners in the community.

ELIGIBILITY:
Inclusion Criteria:

* HIV-diagnosed
* Sexually active (penile-vaginal or penile-anal) and/or sharing injection equipment during the year before incarceration

Exclusion Criteria:

* Incarcerated more than 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
HIV Testing | 6 weeks after randomization
  Number of partners who complete HIV testing

SECONDARY OUTCOMES:
HIV Notification | 6 weeks post-randomization
  Number of partners who are notified of possible shared exposure to HIV
First HIV Test | 6 weeks post-randomization
  Number of partners who are HIV testing for the first time
HIV Diagnosis | 6 weeks post-randomization
  Number of partners who are HIV diagnosed
ART Linkage | 6 weeks post-randomization
  Number of HIV-diagnosed partners who are evaluated for treatment by a physician
ART Initiation | 6 weeks post-randomization
  Number of HIV-diagnosed partners who initiate treatment with antiretroviral therapy (ART)

CONTACTS AND LOCATIONS:
Overall Officials: Agung Waluyo, PhD, Principal Investigator — Indonesia University; Gabriel Culbert, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- Fakultas Ilmu Keperawatan, Universitas Indonesia, Depok, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
All data collected for this study will follow the NIH Policy for Data Management and Sharing (NOT-OD-21-013) and NIMH's extensions that apply to HIV-related applications that involve human subject research funded by NIMH. Raw and analyzed data from this study will be deposited into the NIMH Data Archive (NDA). Other data outputs also will be housed in the University of Illinois Chicago institutional repository, INDIGO, which is able to store non-sensitive information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will share data with the research community when papers using the data have been accepted for publication or at the end of the award period, whichever occurs sooner.
Access Criteria: Access to de-identified scientific data will not be restricted. Due to the sensitive nature of the topic, identifiable data will be limited to sharing through data use agreements.

REFERENCES:
- [Background] Culbert GJ, Levy JA, Steffen AD, Waluyo A, Earnshaw VA, Rahadi A. Impart: findings from a prison-based model of HIV assisted partner notification in Indonesia. J Int AIDS Soc. 2023 Jun;26(6):e26132. doi: 10.1002/jia2.26132. PMID 37339342